CLINICAL TRIAL: NCT07196306
Title: Study of Subcutaneous Sarilumab vs Placebo in Hospitalized Patients With Respiratory Distress Caused by COVID 19
Brief Title: Subcutaneous Sarilumab vs Placebo in Hospitalized Patients With Respiratory Distress Caused by COVID 19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: BayCare Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2020-05-07; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: COVID; COVID-19; Corona Virus Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — sarilumab

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sarilumab (Experimental): 200 mg in 1.14 mL Subcutaneous x 1 or 2 dose(s)
  Interventions: Drug: Sarilumab 200 MG/1.14 ML Subcutaneous Solution
- Placebo (Placebo Comparator): Normal saline 0.9% 1.14 mL Subcutaneous x 1 or 2 dose(s)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sarilumab 200 MG/1.14 ML Subcutaneous Solution — At the time of enrollment, the intervention arm subjects are administered single or double dose of study drug while the placebo arm subjects are administered the placebo drug (normal saline). Subjects will be assigned to the intervention or placebo arm in random order.
  Arms: Sarilumab
Drug: Placebo — Normal saline 0.9% 1.14 mL Subcutaneous x 1 or 2 dose(s)
  Arms: Placebo

SUMMARY:
Studying the efficacy of IL-6 inhibition utilizing single or double dose subcutaneous administration of Sarilumab in patients with severe respiratory distress caused by COVID19 regarding improvement in oxygen demands and other clinical outcomes.

DETAILED DESCRIPTION:
At the time of writing this protocol, there does not exist any strategy to treat acute respiratory distress syndrome associated with COVID-19. Due to the overwhelming health crisis facing a large portion of the population, and due to lack of standardization or clinical approach to management of severe respiratory failure short of standard of care with oxygenation and supportive measures, we elected to embark on this study to evaluate the role of IL-6 stimulating the immune system and the effect of inhibiting signal propagation on clinical outcome.

For this study, Sarilumab, an FDA approved IL-6 receptor antagonist, currently used for severe rheumatoid arthritis, has been selected. The dose and administration of therapy used for the study conforms to the current FDA recommendation for the primary use of Sarilumab.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed COVID-19 via centralized RT-PCR testing for SARS-CoV2 infection performed at BayCare Health System Laboratory or associated and accredited laboratory.
2. Subjects must be hospitalized.
3. Document fever of 100.4 F or more during hospitalization and prior to enrollment.
4. Evidence of abnormal chest imaging chest x-ray or CT.
5. Moderate to severe respiratory distress requiring oxygen supplementation as defined by criteria listed below.

   "Oxygen saturation (Sao2) of 92% or less on room air or a ratio of the partial pressure of oxygen (Pao2) to the fraction of inspired oxygen (Fio2) of less than 200 mm Hg, on ventilator settings that include PEEP ≥5 cm H2O".
6. Subjects may have active co-infection with other respiratory pathogens.
7. Males and non-pregnant females at least 18 years of age.

Exclusion Criteria:

1. The subject or Legally Authorized Representative is unable to provide consent in person or by phone.
2. The subject is participating in any other clinical trial for treatment of COVID 19 or any other treatment related clinical trial for a concurrent disease. No plans for additional COVID trials.
3. The subject does not meet criteria for moderate to severe respiratory distress.
4. The presence of any of the following lab abnormalities. ANC <2000/mm3, Platelet count <50,000/mm3, ALT/AST >6x ULN
5. Prior utilization of any IL-6 inhibitors or receptor antagonists at any time in patient's life, JAK inhibitors, DMARDS(Except Hydroxychloroquine), long term, chronic steroid use (more than 6 months) or mTOR inhibitors.
6. The subject has history of organ or bone marrow transplant.
7. History of active or incompletely treated Tuberculosis (TB).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Time to clinical outcome improvement | Time to improvement up to 28 days
  Time from randomization to improvement in oxygenation. Improvement in oxygenation is defined as SpO2/FiO2 improvement by 100 or greater.

SECONDARY OUTCOMES:
Time to improvement in oxygenation | Time to improvement up to 28 days
  Time from randomization to no requirement of any oxygen supplementation with Oxygen saturation of > =92% at rest.
The number of patients with a need for intubation | Up to 28 days
Time on ventilator | Up to 28 days
Fever resolution | Up to 28 days
  A continuous period at least 48 hours without a recorded temperature equal or more than 100.4 F.
Hemodynamic improvement to normal range | Up to 28 days
  Heart rate
Improvement or normalization in CBC | At 48 hours post intervention up to 28 days
  CBC with differential
Time to objective improvement noted on chest imaging | Up to 28 days
Time from randomization to hospital discharge | Up to 28 days
Death | Up to 28 days
Hemodynamic improvement to normal range | Up to 28 days
  Respiratory rate
Improvement or normalization in CMP | At 48 hours post intervention up to 28 days
  Comprehensive Metabolic Panel
Improvement or normalization in LDH | At 48 hours post intervention up to 28 days
  LDH
Improvement or normalization in Lactic Acid | At 48 hours post intervention up to 28 days
  Lactic Acid
Improvement or normalization in Procalcitonin | At 48 hours post intervention up to 28 days
  Procalcitonin
Improvement or normalization in Ferritin | At 48 hours post intervention up to 28 days
  Ferritin
Improvement or normalization in CRP | At 48 hours post intervention up to 28 days
  CRP
Improvement or normalization in D-Dimer | At 48 hours post intervention up to 28 days
  D-Dimer
Improvement or normalization in IL-6 | At 48 hours post intervention up to 28 days
  IL-6

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Mauck, BA, Study Director — BayCare Health System
Locations (3):
- United States (3):
  - Morton Plant Hospital, Clearwater, Florida
  - St. Anthony's Hospital, St. Petersburg, Florida
  - St. Joseph's Hospital, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No